CLINICAL TRIAL: NCT02920931
Title: A Randomized, Open-label, Single-dosing, 2X2 Crossover Study to Compare the Safety and Pharmacokinetics of BR-TND Tablet(Tenofovir Disoproxil) With Viread Tablet(Tenofovir Disoproxil Fumarate) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-TND-CT-101
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-12

CONDITIONS: Hepatitis
MeSH Terms: conditions — Hepatitis | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 1. st period: Tenofovir disoproxil fumarate
  2. nd period: Tenofovir Disoproxil
  Interventions: Drug: Tenofovir disoproxil
- B (Active Comparator): 1. st period: Tenofovir disoproxil
  2. nd period: Tenofovir Disoproxil fumarate
  Interventions: Drug: Tenofovir disoproxil

INTERVENTIONS:
Drug: Tenofovir disoproxil

SUMMARY:
A Randomized, Open-label, Single-dosing, 2X2 Crossover Study to Compare the Safety and Pharmacokinetics of BR-TND Tablet(Tenofovir Disoproxil) With Viread Tablet(Tenofovir Disoproxil Fumarate) in Healthy Male Volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject, aged 19- 45 years at screening.
2. Body weight of ≥ 55 kg and within ± 20% of ideal body weight (IBW)(kg) = {height (cm) - 100} * 0.9
3. No morbid symptom or sign, based on physical examination, with no innate or chronic disease.
4. Subject that is considered appropriate for participating in the study by an investigator, based on clinical laboratory test (hematology, clinical chemistry, urinalysis) that is performed according to the characteristics of investigational drugs.
5. Subjects must be able to listen to and understand the detailed statement of informed consent, and willing to decide to participate in the study, follow the study directions and provide written informed consent.

Exclusion Criteria:

1. A clinically significant disease or history in hepatobiliary system, kidney, digestive system, respiratory system, hemato-oncological system, endocrine system, neuro-psychiatric system, musculo-skeletal system, immune system, otorhinolaryngological system or cardiovascular system.
2. A history of gastrointestinal system disorder(i.e, Crohn's disease, ulcer, acute or chronic pancreatitis) or surgery (excluding simple appendectomy or herniorrhaphy) that may affect absorption of investigational drugs.
3. A history of hypersensitivity to investigational drugs and its additives or clinically significant hypersensitivity to any other drug.
4. Galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption and any other hereditary disorder.
5. Vital sign measured in sitting position meets any one of following results; systolic blood pressure > 140 mmHg or <100 mmHg, diastolic blood pressure > 90 mmHg or <60 mmHg, pulse ≥ 100 times/min.
6. Aspartate aminotransferase(AST) or Alanine aminotransaminase(ALT) > 2 times upper normal limit, or Total bilirubin > 2 times upper normal limit.
7. Renal disorder (Creatinine clearance < 50 mL/min, calculated by Cockcroft-Gault formula)
8. Positive in serologic tests (RPR Ab(VDRL), HBsAg, hepatitis C virus (HCV) Ab, anti HIV(AIDS))
9. History of drug abuse, or positive in drug screening test.
10. Use of inducer or inhibitor of metabolic enzymes for drugs like barbiturate.
11. Use of any prescribed drugs or herbal remedies within 2 weeks, or use of any over-the-counter medication within 1 week prior to the first administration of investigational drug, and this will affect this study or the safety of the subjects at discretion of study investigator.
12. Participation in another clinical trial or a bioequivalent study within 3 months prior to the first administration of investigational drug (The finish time of previous study is the day of the last administration of study drug)
13. Whole blood donation within 2 months or component donation within 1 month, prior to the first administration of investigational drug, or transfusion within 1 month prior to the first administration of investigational drug.
14. Prolonged excessive alcohol consumption (>21 units/week, 1 unit=10g of pure alcohol), or subjects who can not abstain from drinking from 24 hours prior to hospitalization until the discharge.
15. Smoking more than 10 cigarettes per day, excessive caffeine consumption (example: instant coffee > 5 cups/day)
16. Subjects planning to get a dental treatment(tooth extraction, orthodontic treatment, endodontic treatment etc) and a selective surgery(aesthetic surgery, LASIK, LASEK etc) during the period from informed consent form(ICF) to post-study visit, which is impossible to be postponed.
17. Subjects who are judged to be inappropriate for this study by investigators according to other reasons including clinical lab test result

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration(Cmax) of Tenofovir | 0~72 hour after medication
Area under the curve(AUCt) of Tenofovir | 0~72 hour after medication

CONTACTS AND LOCATIONS:
Overall Officials: Jang Hee Hong, PhD, Principal Investigator — Chungnam National University
Locations (1):
- ChungNam university hospital, Jungnam, South Korea

IPD SHARING:
Plan to Share IPD: No